CLINICAL TRIAL: NCT00873769
Title: Pharmacokinetics of Staccato® Loxapine for Inhalation in Smokers Compared to Nonsmokers
Brief Title: Staccato Loxapine PK in Smokers and Nonsmokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMDC-004-106; 27 February 2009
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2009-06

CONDITIONS: Smoking, Cigarette
Keywords: Staccato Loxapine; pharmacokinetics; smokers; non-smokers
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Masking Description: Single-center, single-dose, single-treatment, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy smokers (Experimental): Healthy smokers, male and female
  Interventions: Drug: Inhaled Loxapine 10 mg
- Healthy nonsmokers (Experimental): Healthy nonsmokers, Healthy smokers, male and female
  Interventions: Drug: Inhaled Loxapine 10 mg

INTERVENTIONS:
Drug: Inhaled Loxapine 10 mg — Staccato Loxapine 10 mg, single dose
  Other Names: Staccato Loxapine 10 mg

SUMMARY:
The objective of this trial was to assess the pharmacokinetics of a single dose of 10 mg Staccato Loxapine administered to smokers compared to nonsmokers.

DETAILED DESCRIPTION:
Pharmacokinetics and sedation pharmacodynamics were studied using a visual analog scale were studied in male and female adult subjects (nonsmokers and smokers) following a single dose of 10 mg of inhaled loxapine. Blood samples were drawn at predose, 30 seconds, 1, 2, 3, 10, 30, and 60 minutes, and 2, 6, 12, and 24 hours after dosing. Loxapine and 8-OH-loxapine were analyzed using reverse-phase liquid chromatography coupled with a tandem mass spectrometer.

ELIGIBILITY:
Inclusion Criteria:

* Normal spirometry at screening and in good general health as determined by a complete medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, and urinalysis,
* Smokers must have a history of smoking > 15 cigarettes/day currently and for at least the last 2 years,
* Nonsmokers must have never smoked > 5 cigarettes/day and not smoking at all for at least the last 2 years.

Exclusion Criteria:

* Any acute illness in the 5 days,
* Use of a bronchodilator for the treatment of wheezing within 12 months, OR
* Any other disease or condition, by history, physical examination, or laboratory abnormalities that would present undue risk to the subject, or may confound the interpretation of study results.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Noncompartmental Pharmacokinetic parameters | 24 hours

SECONDARY OUTCOMES:
Vital signs | 24 hours
Treatment emergent adverse events | 24 hours
Sedation visual analog scale | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Randall R. Stoltz, MD, Principal Investigator — Covance Clincial Research Unit, Inc.
Locations (1):
- Covance Clinical Research Unit, Inc., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Takahashi LH, Huie K, Spyker DA, Fishman RS, Cassella JV. Effect of smoking on the pharmacokinetics of inhaled loxapine. Ther Drug Monit. 2014 Oct;36(5):618-23. doi: 10.1097/FTD.0000000000000048. PMID 24937085